CLINICAL TRIAL: NCT00905528
Title: Prospective Study on Endothelial Function in Subjects With Type 2 Diabetes Mellitus
Brief Title: TRENDY Follow-up: Study on Endothelial Function in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: Re.-No. 3204; SFB TP B5
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; endothelial function; renal hemodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Telmisartan; Ramipril

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Subjects with type 2 diabetes mellitus, eGFR > 80, hypertension, no overt proteinuria
  Interventions: Drug: Telmisartan 80 mg/d
- B: Subjects with type 2 diabetes mellitus, eGFR > 80, hypertension, no overt proteinuria
  Interventions: Drug: Ramipril 10 mg/d

INTERVENTIONS:
Drug: Telmisartan 80 mg/d
  Groups: A
Drug: Ramipril 10 mg/d
  Groups: B

SUMMARY:
Basal nitric oxide (NO) activity plays a pivotal role in the regulation of glomerular hemodynamics, and in animal experiments its alteration has been associated with morphological changes characteristic of diabetic nephropathy. The investigators aimed to assess in a prospective study: 1. basal NO activity of renal vasculature and 2. renal hemodynamics to examine whether impairment of basal NO activity of the renal vasculature is related to development and progression of diabetic nephropathy and other cardiovascular endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus

Exclusion Criteria:

* Macroalbuminuria
* Symptomatic cardiovascular disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 2 diabetes mellitus and normo or microalbuminuria
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2002-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change in eGFR after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, Prof., Principal Investigator — Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Ritt M, Ott C, Delles C, Schneider MP, Schmieder RE. Impact of the endothelial nitric oxide synthase gene G894T polymorphism on renal endothelial function in patients with type 2 diabetes. Pharmacogenet Genomics. 2008 Aug;18(8):699-707. doi: 10.1097/FPC.0b013e32830500b1. PMID 18622262
- [Result] Ritt M, Ott C, Raff U, Schneider MP, Schuster I, Hilgers KF, Schlaich MP, Schmieder RE. Renal vascular endothelial function in hypertensive patients with type 2 diabetes mellitus. Am J Kidney Dis. 2009 Feb;53(2):281-9. doi: 10.1053/j.ajkd.2008.10.041. Epub 2008 Dec 19. PMID 19100670
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786